CLINICAL TRIAL: NCT05637567
Title: Perioperative Platelet Inhibition With Acetylsalicylic Acid Targeting Intraoperative Tumor Cell Seeding in Patients With Resectable Tumors of the Pancreatic Head - a Randomized, Controlled Multicenter Study
Brief Title: Perioperative Platelet Inhibition With Acetylsalicylic Acid in Patients With Resectable Tumors of the Pancreatic Head
Acronym: ASAP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DKFZ-2022-006
Record Dates: First submitted 2022-11-24; First posted 2022-12-05 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Pancreatic Cancer Resectable
Keywords: pancreatic cancer; pancreatic head cancer; acetylsalicylic acid; aspirin; pancreatic head resection; liver metastases; distant metastases; circulating tumor cells
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplastic Cells, Circulating | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): 100 mg acetylsalicylic acid per os once daily, starting 1-4 weeks before surgery until 6 months after surgery
  Interventions: Drug: Acetylsalicylic acid
- Control Arm (Placebo Comparator): Identically looking placebo pill, starting 1-4 weeks before surgery until 6 months after surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetylsalicylic acid — 100 mg per os once daily
  Arms: Treatment Arm
Drug: Placebo — Placebo pill per os once daily
  Arms: Control Arm

SUMMARY:
This randomized, controlled clinical trial compares the perioperative treatment with acetylsalicylic acid (aspirin) in patients with cancer of the pancreatic head. The main question it aims to answer is: Do patients treated perioperatively with aspirin develop less metastasis after curative resection of pancreatic head tumors?

Participants will be asked to :

* take a daily aspirin tablet starting 1-4 weeks before surgery until 6 months after surgery
* participate in regular follow-up visits.

DETAILED DESCRIPTION:
With few symptoms, rapid progression and early metastasis pancreatic cancer (pancreatic ductal adenocarcinoma, PDAC) is the third leading cause of cancer death worldwide. In early stages of PDAC, surgical resection followed by adjuvant chemotherapy is the mainstay of treatment. Unfortunately, the majority of patients develop tumor recurrence (most frequently in the liver) despite complete resection and adjuvant treatment. This early postoperative recurrence is a result of preoperatively present, undetected micrometastases, and, most importantly, iatrogenic dissemination of circulating tumor cells (CTCs) by surgical manipulation of the tumor during resection. CTCs can be detected in the majority of PDAC patients and correlate with worse overall survival.

Survival of CTCs in the hostile environment of circulation requires resistance to physical forces (i.e., turbulence, shear stress), but also immune escape mechanisms to avoid clearance by immune cells such as natural killer (NK) cells. CTCs are highly heterogeneous and, by the majority, non-tumorigenic. The number of other nucleated blood cells such as leukocytes greatly exceeds the number of CTCs; in many solid tumors including PDAC, the average number of (detectable) CTCs is less than 10 cells / mL of whole blood. This demonstrates the inefficiency of the metastatic process, which is at least partially a result of early clearance of CTCs after entering the blood stream.

After entering circulation, the first cells that CTCs come in direct contact with are platelets. This leads to activation of platelets and aggregation on the CTCs, which are thus enveloped and protected from the hostile environment in the circulation. This effect is seen in many, but not all CTCs, the underlying molecular mechanisms are currently being investigated. It is conceivable that not only shear forces and turbulence have less influence on CTCs enveloped by platelets, but also that immune cells (e.g. NK cells) in the bloodstream are less likely to detect and eliminate CTCs and therapeutic antibodies have fewer binding sites.

Arguably the most decisive days in the lives of cancer patients are when they undergo surgery for tumor resection. For most solid tumors, surgery is part of all curative treatment regimens. However, the occurrence of distant metastases often brings surgery to its limits, either because not all metastatic lesions are resectable, or due to rapidly recurring metastatic disease after surgery. Many patients develop disseminated disease early after curative resection of an initially non-metastatic tumor. There are several potential reasons behind this phenomenon, most prominently the immunosuppression resulting from major surgery and the iatrogenic dissemination of CTCs during surgery. Surgery-related immunosuppression is addressed by continuous improvement of perioperative medicine such as prehabilitation or early recovery / fast-track programs as well as minimally invasive surgical procedures, whenever possible. However, only few measures have been taken so far to reduce iatrogenic dissemination of tumor cells during PDAC surgery.

During cancer surgery, the tumor is inevitably touched, manipulated or even squeezed as it has to be mobilized from its surroundings while limiting the damage to neighboring structures. This manipulation of the tumor leads to iatrogenic CTC dissemination. The only clinically used measure to reduce tumor cell dissemination during surgery is currently an early ligation of tumor-draining veins prior to manipulation and mobilization of the tumor mass. This method can only be employed in tumor entities that are drained by one or few well-defined veins such as lung cancer or colorectal cancer, in which this method is successfully applied. In other tumors, which are drained by multiple small and/or initially inaccessible vessels (e.g., hepatic tumors) or in which the tumor-draining vein cannot be occluded for prolonged periods of time (e.g., the portal vein draining tumors of the pancreatic head), this "vein first" or "no touch" approach is not applicable. Since especially in pancreatic tumors, hepatic recurrence often occurs after curative resection and inevitably leads to the death of the patient, this represents a major clinical problem.

Approximately 5% of cancer patients are on permanent medication with platelet inhibition (PI), most prominently acetylsalicylic acid (ASA, aspirin) for a cardiac indication. ASA is usually taken orally at a dosage of 100 mg once a day and several studies and meta-analyses have shown that perioperative ASA intake at this standard dosage leads only to a slightly increased risk of bleeding. Therefore, platelet aggregation inhibition with aspirin alone is continued perioperatively nowadays and is classified as safe.

ASA medication leads to increased overall survival in several cancer entities. A meta-analysis of 22 studies evaluating survival of colorectal cancer patients in dependence of ASA treatment revealed a significant survival advantage for patients with continuous ASA treatment in comparison with patients who did not take ASA or terminated ASA intake prior to or at the time point of tumor diagnosis.

So far, despite ample preclinical evidence, only few clinical studies have investigated the effect of ASA treatment on PDAC. Recently published, retrospective data indicates a significantly improved survival after curative resection of PDAC for patients with perioperative low-dose ASA medication, which is directly attributable to a reduced postoperative incidence of distant metastases. A preliminary meta-analysis (incorporating a second study investigating ASA treatment in PDAC) confirms the significantly improved disease-free survival after resection of PDAC in patients under permanent platelet inhibition with ASA. There is also evidence of a reduced incidence of distant metastases under ASA treatment in other tumor entities.

The investigators hypothesize that the reason for the reduced incidence of distant metastases achieved by ASA is the inhibited platelet-mediated protection of CTCs.

In conclusion, perioperative platelet inhibition with ASA may drastically reduce the postoperative incidence of hematogenous metastases with very low toxicity and risk to the patients with PDAC. Despite this favorable benefit-risk ratio, no prospective, randomized-controlled trials investigating this treatment have been conducted. As a result and despite its potential benefits, perioperative ASA treatment in patients undergoing resection of the pancreatic head for malignant indications is currently not generally recommended.

The aim of this multicentric randomized-controlled trial is therefore to investigate the impact of perioperative ASA treatment on the occurrence of hematogenous metastases, survival and perioperative complications in patients undergoing pancreatic head resection (pylorus-preserving pancreaticoduodenectomy / Traverso-Longmire procedure) for PDAC.

ELIGIBILITY:
Inclusion Criteria:

1. Indication: Patients with (histologically confirmed or clinically suspected) surgically resectable, non-metastatic ductal adenocarcinoma of the pancreatic head
2. Patients planned for pylorus-preserving partial pancreaticoduodenectomy (PPPD / "ppWhipple" / Traverso-Longmire procedure) (conventional or minimally invasive)
3. Male and female patients aged 18 to 80 years
4. Written informed consent of the participating person
5. ECOG≤2

Exclusion Criteria:

1. Metastatic disease (distant or peritoneal metastases or lymph node involvement considered distant metastasis (i.e., interaortocaval nodes))
2. Preoperative use of anticoagulants / thrombolytics (e.g. warfarin, heparin), platelet aggregation inhibitors (e.g. ASA, ticlopidine, clopidogrel), chronic NSAID or metamizole use
3. Neoadjuvant treatment for locally advanced disease
4. Presumed necessity of arterial resection (other than gastroduodenal artery)
5. Advanced liver (INR >1.5 or hepatic encephalopathy) or renal failure (stage IV or higher)
6. Advanced heart disease (NYHA class ≥ 3)
7. Known hypersensitivity to ASA or to drugs with a similar chemical structure
8. History of asthma attacks triggered by salicylates or substances with similar effects
9. Haemorrhagic diathesis, blood coagulation disorders such as haemophilia or thrombocytopenia
10. Thrombocytosis > 450,000 / μL
11. Methotrexate at a dosage of 15 mg or more per week
12. Participation in competing trials affecting the effects of the investigational medicinal product (IMP) or outcome measures
13. Addictive or other medical conditions that do not allow the subject to appreciate the nature and scope of the clinical trial and its potential consequences
14. Pregnant or breast-feeding women
15. Women of childbearing potential, except women who meet the following criteria:

    * Post-menopausal (12 months natural amenorrhoea or six months amenorrhoea with serum follicle-stimulating hormone (FSH) > 40 U/ml)
    * Postoperative (six weeks after bilateral ovariectomy with or without hysterectomy)
    * Regular and correct use of a contraceptive method with a failure rate < 1% per year (e.g. implants, depot injections, oral contraceptives, intrauterine devices)
    * Sexual abstinence
    * Vasectomy of partner
16. Indications that the patient is unlikely to comply with the protocol (e.g. unwillingness to cooperate)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Hematogenous metastases-free survival | 24 months
  The primary efficacy endpoint of the study is hematogenous metastases-free survival (HMFS), which is defined as the time from the day of surgery to the date of diagnosis of hematogenous distant metastases (e.g., hepatic or pulmonary metastases) or date of death from any cause, whichever comes first. Peritoneal metastases (peritoneal carcinomatosis) are not regarded hematogenous metastases. The HMFS status is evaluated at regular follow-up examinations for 36 months postoperatively and further recorded during clinical follow-up visits until the end of the trial.

SECONDARY OUTCOMES:
Overall survival | 24 months
  Overall survival (OS) is defined as the time from the day of surgery until death from any cause.
Cancer-specific survival | 24 months
  Cancer-specific survival (CSS) is defined as the time from the day of surgery until death due to the treated cancer or a treatment-related complication.
Disease-free survival | 24 months
  Disease-free survival (DFS) is defined as the time from the day of surgery to the date of diagnosis of tumor recurrence (in any location) or to the date of death from any cause, whichever comes first.
Intraoperative blood loss | During surgery
  Intraoperative blood loss is documented in milliliters during surgery and subsequently analyzed. Intraoperative transfusions of blood or blood components will also be recorded and analyzed.
Duration of surgery | During surgery
  The duration of surgery (first incision to wound closure) is recorded and subsequently analyzed.
Perioperative surgical complications | Until 90 days after surgery
  Surgical complications include postoperative bleeding, anastomotic insufficiencies, pancreatic fistulas, wound infections, fascial dehiscence, delayed gastric emptying (DGE) and gastrointestinal atony.
Perioperative medical complications | Until 90 days after surgery
  Medical complications include pneumonia, myocardial infarction, cardiac decompensation, new onset atrial fibrillation, respiratory insufficiency, renal failure, liver failure and sepsis. Other complications include allergic or intolerance reactions, cerebral infarctions, delirium and pain, prolonging the length of hospital stay.
R status | during surgery
  Will be recorded from pathology report.
Number of resected lymph nodes | during surgery
  Will be recorded from pathology report.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Schoelch, MD, Study Chair — German Cancer Research Center

IPD SHARING:
Plan to Share IPD: No